CLINICAL TRIAL: NCT01984528
Title: Biological Standardization of Alternaria Alternata Allergen Extract to Determine the Biological Activity in Histamine Equivalent Units (HEP).
Brief Title: To Determine the Minimum Amount of Alternaria Alternata Allergen Extract Producing a Positive Skin Reaction.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 301-PR-PRI-198; 2013-001308-13 (EudraCT Number)
Record Dates: First submitted 2013-11-08; First posted 2013-11-14 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2013-05

CONDITIONS: Allergy to Alternaria Fungus
Keywords: Immunotherapy; Skin prick test; Standardization; Alternaria alternata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prick Test (Experimental): Alternaria alternata allergen extract Positve control Negative control
  Interventions: Biological: four differente concentrations of Alternaria alternata allergen extract, positive control and negative control

INTERVENTIONS:
Biological: four differente concentrations of Alternaria alternata allergen extract, positive control and negative control — This concentrations will be tested in every patient in duplicate on the volar surface of the forearm.
  Other Names: Four concentratios of Alternaria alternata together with a positive and negative control.

SUMMARY:
The objetive of this study is to determine the minimum amount of Alternaria alternata allergen extract producing in a positive skin reaction.

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. The primary objective is to assess the concentration of alternaria alternata allergen extract that elicits a wheal size equivalent to that of a 10 mg/ml histamine dyhidrochloride solution.

ELIGIBILITY:
Inclusion Criteria:

Positive clinical history of inhalatory allergy to Alternaria alternata. Subject has provided written informed consent, appropriately signed and dated by the subject.

Subject can be male or female of any race and ethnic group. -Age > and =18 years and < and = 60 years at the study inclusion day.

Positive skin prick test with a standardized commercially available preparation of Alternaria alternata allergen extract. The skin prick test will be considered positive if the test results in a wheal major diameter of at least 3 mm or wheal area ≥ 7 mm2. Positive skin prick test results are valid if performed within one year prior to the inclusion of the subject in the study.

A positive test for specific IgE to alternaria alternata (CAP-RAST major or equal to 2). IgE results are valid if performed within one year prior to the inclusion of the subject in the study.

The mean wheal diameters of the obtained with histamine dihydrochloride (10 mg / ml) in the forearm ≥ 3 mm.

Exclusion Criteria:

Immunotherapy in the past 5 years with an allergen preparation known to interfere with the allergen to be tested (for example: fungal extracts) Use of drugs that may interfere with the skin reactions (e.g., antihistamines). Treatment with any of the following medications: oral tricyclic or tetracyclic antidepressants, beta-blockers, corticosteroids (major 10 mg/daily of prednisone or equivalent).

Women who are pregnant or breastfeeding period and women with positive pregnancy test at Visit 1 or 2.

Dermographism affecting the skin area at the test site at either study visit. Atopic dermatitis affecting the skin area at the test site at either study visit.

Urticaria affecting the skin area at the test site at either study visit. Diseases of the immune system relevant clinically, both autoimmune and immunodeficiencies.

Serious diseases not controlled that may increase the risk for the safety of the subjects involved in this study, including, but not limited to the following: heart failure, uncontrolled or severe respiratory diseases, endocrine diseases, clinically relevant kidney or liver diseases or hematological diseases.

Participation in any other clinical trial within 30 days prior to the inclusion of the subject in this clinical trial. Patients with diseases or conditions that limit the use of adrenaline (heart disease, severe hypertension).

Severe psychiatric, psychological or neurological disorders. Abuse of alcohol, drugs or medicines in the previous year. Subjects who have received anti-IgE (Omalizumab).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) on the skin at the site of the puncture during the immediate phase. | Test sited chould be inspected and recorded 15-20 min after appliction

CONTACTS AND LOCATIONS:
Overall Officials: Lena Erbiti, Study Chair — Laboratorios Leti, S.L.U; Santiago Quirce, MD, Principal Investigator — Hospital Universitario La Paz; José Damian López, MD, Principal Investigator — HOSPITAL CLÍNICO UNIVERSITARIO VIRGEN DE LA
Locations (2):
- Spain (2):
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Clínico Universitario Virgen de La Arrixaca, El Palmar, Murcia